CLINICAL TRIAL: NCT03522441
Title: A Multi-Center, Double-Blind, Randomized, Vehicle-Controlled, Parallel-Group Study Comparing Clindamycin 1% Gel To Clindamycin 1% Gel (Greenstone LLC) and Both Active Treatments to Vehicle Control in the Treatment of Acne Vulgaris
Brief Title: Bioequivalence Study of Clindamycin Gel 1% in Treatment of Acne Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Akorn, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLMG 1711
Record Dates: First submitted 2018-04-23; First posted 2018-05-11 (Actual); Results first posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2018-05

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Clindamycin; Gels

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Clindamycin 1% gel (Akorn Pharmaceuticals) (Experimental)
  Interventions: Drug: Clindamycin 1% Gel
- Clindamycin 1% gel (Greenstone LLC) (Active Comparator)
  Interventions: Drug: Clindamycin 1% Gel
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clindamycin 1% Gel — Topical gel
  Arms: Clindamycin 1% gel (Akorn Pharmaceuticals); Clindamycin 1% gel (Greenstone LLC)
Drug: Placebo — Topical Placebo gel
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, multiple-site, placebo-controlled, parallel-group study, designed to compare the efficacy and safety of generic Clindamycin 1% gel (Akorn), and the marketed product Clindamycin 1% gel (Greenstone LLC) in the treatment of acne vulgaris.

ELIGIBILITY:
IInclusion Criteria:

* Male or non-pregnant, non-lactating female, ≥12 and ≤40 years of age with a clinical diagnosis of acne vulgaris.
* Have facial acne with: ≥20 facial inflammatory lesions (papules and pustules) and ≥25 non-inflammatory lesions (open and closed comedones), and ≤2 nodulocystic lesions (nodules and cysts) and have an IGA score of 2, 3 or 4.

Exclusion Criteria:

* Subject has more than 2 facial nodular lesions; any nodules present will be documented but not included in the inflammatory lesion count for analysis.
* Subject has active cystic acne.
* Subject has acne conglobata.
* Subjects with excessive facial hair such as beards, sideburns, moustaches, etc. that would interfere with the diagnosis or assessment of acne.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1125 (Actual)
Dates: Start 2018-04-27 (Actual); Primary Completion 2019-04-22 (Actual); Study Completion 2019-04-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (10):
  - Site 11, Encino, California
  - Site 10, Sherman Oaks, California
  - Site 1, Brandon, Florida
  - Site 4, Miramar, Florida
  - Site 5, Miramar, Florida
  - Site 2, Tampa, Florida
  - Site 3, Tampa, Florida
  - Site 12, High Point, North Carolina
  - Site 8, El Paso, Texas
  - Site 9, El Paso, Texas
- Belize (2):
  - Site 6, Belize City
  - Site 7, Belize City

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Clindamycin 1% Gel (Akorn Pharmaceuticals) | Clindamycin 1% Gel (Greenstone LLC) | Placebo
Started | 450 | 450 | 225
Completed | 424 | 431 | 214
Not Completed | 26 | 19 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clindamycin 1% Gel (Akorn Pharmaceuticals) | Clindamycin 1% Gel (Greenstone LLC) | Placebo | Total
Number analyzed (Participants) | 450 | 450 | 225 | 1125
Age, Continuous [Mean (Standard Deviation); unit: year] | 21.3 (7.38) | 20.6 (6.79) | 21.3 (7.01) | 21.0 (7.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 163 | 177 | 88 | 428
  Male | 287 | 273 | 137 | 697
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 7 | 1 | 1 | 9
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 173 | 170 | 73 | 416
  White | 264 | 274 | 148 | 686
  More than one race | 5 | 5 | 3 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in the Number of Inflamed Lesions (Papules/Pustules)- Time Frame: Baseline to 12 Weeks
Time Frame: Percent change from baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: % mean change from baseline
Arm/Group | Clindamycin 1% Gel (Akorn Pharmaceuticals) | Clindamycin 1% Gel (Greenstone LLC) | Placebo
Number analyzed (Participants) | 424 | 431 | 214
% mean change from baseline | -66.22 (28.002) | -72 (27.19) | -16.02 (34.238)

2. Primary Outcome: Percent Change in the Non-inflammatory (Open and Closed Comedones) Lesion Counts - Change in Baseline to 12 Week
Time Frame: Percent change in baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Clindamycin 1% Gel (Akorn Pharmaceuticals) | Clindamycin 1% Gel (Greenstone LLC) | Placebo
Number analyzed (Participants) | 424 | 431 | 214
percent change from baseline | -50.45 (29.934) | -57.42 (25.709) | -46.07 (29.922)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Clindamycin 1% Gel (Akorn Pharmaceuticals) | Clindamycin 1% Gel (Greenstone LLC) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/450 | 0/450 | 0/225
Serious Adverse Events (participants affected / at risk) | 0/450 | 0/450 | 0/225
Other Adverse Events (participants affected / at risk) | 0/450 | 0/450 | 0/225

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-23): https://cdn.clinicaltrials.gov/large-docs/41/NCT03522441/Prot_SAP_002.pdf